CLINICAL TRIAL: NCT00781820
Title: A Double-blind, Randomized, Multicenter, Placebo- Controlled Phase 3 Trial to Prove the Superiority of Bifonazole vs. Placebo After 4 Weeks of Onychomycosis Treatment/ as a Follow-up of a 2 Weeks Treatment of Non-surgical Nail Ablation of Diseased Nail Matrix With 40% Urea Paste
Brief Title: Comparative Efficacy of Bifonazole Cream vs Placebo After Nail Ablation With Urea Paste
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Consumer Care Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12999; 2008-003215-13 (EudraCT Number)
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Onychomycosis
Keywords: Bifonazole; Placebo; Urea; Nail fungus
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo cream
- Arm 1 (Experimental)
  Interventions: Drug: Bifonazole cream 1%

INTERVENTIONS:
Drug: Bifonazole cream 1% — 1 squeeze of Bifonazole cream sufficient to cover the infected nail bed(s) with a thin layer once daily for 28 days after nail ablation with urea paste
  Arms: Arm 1
Drug: Placebo cream — 1 squeeze of Placebo cream sufficient to cover the infected nail bed(s) with a thin layer once daily for 28 days after nail ablation with urea paste
  Arms: Arm 2

SUMMARY:
The study is focused to prove that the efficacy of a 1% Bifonazole cream is superior to a placebo cream after non-surgical nail ablation with a 40% urea paste.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 years;
* Positive clinical findings of onychomycosis according to the judgement of the investigator (e.g. thickening, discoloration, structural changes, misshaped nails);
* Positive mycological findings (positive microscopy and positive culture with identification of pathogen) in material taken from affected nail sites before the start of treatment;
* Nail mycosis with an affected nail area between 20% and 50% in the target nail,
* Nail mycosis in not more than 3 nails (each nail not more than 50% infected area)

Exclusion Criteria:

* Doubtful or negative mycological findings;
* Proximal subungual onychomycosis (PSO);
* Topical antimycotic treatment of feet or hands within 4 weeks prior to screening, topical treatment of onychomycosis of feet or hands within 12 weeks prior to screening;
* Systemic antimycotic treatment within 12 weeks prior to screening;
* Failure to treat tinea pedis/manus (diagnosed at screening) successfully with topical treatment between screening visit and visit 1 (baseline);
* Tinea pedis/manus at visit 1 (baseline);
* Uncontrolled diabetes mellitus
* Psoriasis
* Peripheral arterial disease
* Chronic venous insufficiency;
* Diabetic neuropathy;
* History of hypersensitivity to bifonazole, or any other similar pharmacological agents or components of the products;
* Known sensitivity to plasters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 693 (Actual)
Dates: Start 2008-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Overall cure rate comprising clinical cure and mycological cure microscopy + culture negative | 14 days after end of treatment (=visit 3)

SECONDARY OUTCOMES:
Clinical cure rate | 14 days, 3 and 6 months after end of treatment (=visit 3, 4, and 5)
Culture negative | 14 days, 3 and 6 months after end of treatment (=visit 3, 4, and 5)
Microscopy negative | 14 days, 3 and 6 months after end of treatment (=visit 3, 4, and 5)
Relapse rate (overall cure at visit 3 but positive clinical or mycological findings at visit 4 | 3 and 6 months after end of treatment (=visit 4 and 5)
Mycological cure rate (microscopy + culture negative) | 3 and 6 months after end of treatment (=visit 4 and 5)
Culture negative | 6 months after end of treatment (=visit 5)
Incidence of adverse events | 2 weeks, 3 and 6 months after end of treatment (=visit 3, 4, and 5)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (38):
- Czechia (10):
  - Chomutov
  - Hlinsko
  - Kutná Hora
  - Louny
  - Olomouc
  - Prague
  - Rychnov nad Kněžnou
  - Slaný
  - Svitavy
  - Ústí nad Labem
- Germany (23):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Augsburg, Bavaria
  - Murnau am Staffelsee, Bavaria
  - Oberschleißheim, Bavaria
  - Straubing, Bavaria
  - Potsdam, Brandenburg
  - Hamburg, Hamburg
  - Frankenberg, Hesse
  - Marburg, Hesse
  - Hanover, Lower Saxony
  - Northeim, Lower Saxony
  - Aachen, North Rhine-Westphalia
  - Dülmen, North Rhine-Westphalia
  - Wuppertal, North Rhine-Westphalia
  - Chemnitz, Saxony
  - Dresden, Saxony
  - Leipzig, Saxony
  - Löbau, Saxony
  - Reichenbach, Saxony
  - Halle, Saxony-Anhalt
  - Lübeck, Schleswig-Holstein
  - Berlin, State of Berlin
  - Gera, Thuringia
- Poland (5):
  - Bialystok
  - Gdansk
  - Olsztyn
  - Pruszków
  - Wroclaw